CLINICAL TRIAL: NCT02961634
Title: Study Efficacy and Safety in Comparative Use of Investigational Product Adjuvant Treatment in Onychomycosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: MIP Brasil Indústria e Comércio de Produtos Farmacêuticos LTDA (Industry)
Collaborators: Buranello e Rodrigues Consultoria em Desenvolvimento Farmacêutico Ltda ME (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EN16-0467-01
Record Dates: First submitted 2016-11-07; First posted 2016-11-11 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Onychomycosis
Keywords: onychomycosis; nail
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nailner 2 in 1 + Ciclopirox 8% (Experimental): Patients should apply Nailner 2 in 1 daily in the affected nail 2X a day, morning and night for 30 days. After 30 days passed to apply only 1x daily. No need to sand the nail before the application and the product should be applied on the entire nail, including the sides and the area affected by ringworm. Avoiding wett the nail after application and expose the nail.
  They should also apply ciclopirox 8% nail polish in the first month of treatment every other day (day in and day out). In the second month applied twice a week. In the third month applied once a week. Apply on the affected nails, previously sanded. On the application of two products, Ciclopirox should be applied between the investigational product applications, e.g., in the middle of the day and the investigational product at the beginning and end of the day in the sun.
  Interventions: Device: Nailner 2 in 1; Drug: Ciclopirox 8%
- Ciclopirox 8% (Active Comparator): Patients should also apply ciclopirox 8% nail polish in the first month of treatment every other day (day in and day out). In the second month applied twice a week. In the third month applied once a week. Apply on the affected nails, previously sanded. On the application of two products, Ciclopirox should be applied between the investigational product applications, e.g., in the middle of the day and the investigational product at the beginning and end of the day in the sun.
  Interventions: Drug: Ciclopirox 8%

INTERVENTIONS:
Device: Nailner 2 in 1 — Nailner 2 in 1 is a combination of assets that alter the pH of the nail and is used as an adjunct in the treatment of onychomycosis.
  Arms: Nailner 2 in 1 + Ciclopirox 8%
Drug: Ciclopirox 8% — Ciclopirox 8% is a glaze used in the treatment of onychomycosis

SUMMARY:
Single-center study, single blind, comparative with the objective of evaluating the efficacy and safety of an investigational product as an adjunct in the treatment of onychomycosis improvement of 90 days ± 2 days.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers of both sexes;
* Volunteers aged 18-65 years;
* Volunteers with onychomycosis confirmed by positive direct mycological nail of hands or feet;
* Agreement to comply with the test procedures and attend the clinic in the days and times for certain applications and / or assessments;
* Understand, consent and sign the Instrument of Consent of Clarified.

Exclusion Criteria:

* Pregnancy or risk pregnancy / lactation;
* Use of anti-inflammatory / immunosuppressive drugs (in the last 30 days and during the study);
* Concomitant nail pathologies (psoriasis, lichen planus, etc.);
* Systemic conditions that may compromise the growth of the nail (vascular disease, diabetes, etc.);
* Irritation History to similar products to the investigational product;
* Treatment with antifungal medication prior to the study (up to 12 weeks for systemic medications and topical medications for four weeks);
* Other conditions considered by the investigator physician as reasonable for the disqualification of the individual's participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2017-04 (Estimated); Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Percent of improvement of mycosis by reducing the area of the lesion that will be measured at times D1 and D90 | 90 days
  The improvement rate will be by measuring the area of the nail affected in millimeters (millimeters). The measurement will be taken with a ruler in the direction of the width and length of the lesion (mm2)

SECONDARY OUTCOMES:
Presence of fungal structures in nail affected by onychomycosis in visits 1 and final through mycological examination | 90 days
  Through clinical observation
Number of patients reporting reduction in discomfort caused by onychomycosis through a subjective evaluation questionnaire | 45 and 90 days
  Through the patient's subjective evaluation
Number of adverse events reported and related to the product investigational | 90 days
  Through the spontaneous report of the patients of events occurred during the study

IPD SHARING:
Plan to Share IPD: No